CLINICAL TRIAL: NCT03076359
Title: Traditional Healers as Adherence Partners for PLHIV in Rural Mozambique
Brief Title: Traditional Healers as Adherence Partners for Persons Living With HIV in Rural Mozambique
Acronym: PLHIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Carolyn Audet, Assistant Professor, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 150217; K01MH107255-01 (NIH)
Record Dates: First submitted 2017-03-06; First posted 2017-03-10 (Actual); Results first posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Intervention: This group will receive only standard of care HIV treatment, including ART medications (First-line ART will consist of two nucleoside reverse-transcriptase inhibitors (NRTIs) plus a non-nucleoside reverse-transcriptase inhibitor (NNRTI)- TDF + 3TC (or FTC) + EFV as a fixed-dose combination to be taken twice a day for the rest of the patient's life), clinic-based counseling, and community searches if lost to follow up.
  Interventions: Drug: Standard of Care
- Traditional Healer Support Program (Experimental): This group will receive standard of care as described above. In addition, the investigators will assess an intervention partnership with traditional healer including: community and clinic based support from a trained traditional healer.
  The intervention includes: (1) healer visits to the patient at home, healer support for couples counseling, healer provision of nutritional advice, and healer counsel about the importance of adherence. If anything is amiss, the healer will accompany the patient to the health facility for additional clinical services. In addition, the healer will accompany the patient on all regularly scheduled clinical visits.
  Interventions: Behavioral: Traditional Healer Support Program; Drug: Standard of Care

INTERVENTIONS:
Behavioral: Traditional Healer Support Program — Traditional Healers will provide the "traditional healer support program" assistance, as previously described, to all newly diagnosed patients.
  Other Names: Adherence Support Workers
  Arms: Traditional Healer Support Program
Drug: Standard of Care — First-line ART will consist of two nucleoside reverse-transcriptase inhibitors (NRTIs) plus a non-nucleoside reverse-transcriptase inhibitor (NNRTI)- TDF + 3TC (or FTC) + EFV as a fixed-dose combination to be taken twice a day for the rest of the patient's life), clinic-based counseling, and community searches if lost to follow up.
  Other Names: First Line ART

SUMMARY:
The overall goal of this project is to adapt and assess the impact of a traditional healer training program/intervention on the adherence, retention, and viral load of HIV infected patients newly initiated on anti-retroviral therapy in rural Mozambique.

DETAILED DESCRIPTION:
Incorporating healers as anti-retroviral therapy adherence counselors can help reduce the crisis of HIV treatment abandonment. Healers are often accused of encouraging patients to abandon HIV care, but they can also serve as strong advocates for patient health. When healers were engaged as tuberculosis adherence counselors in South Africa, their patients were as successful as those supported by non-healer counselors. An innovative solution would be to engage trained healers as treatment partners to support medication and appointment adherence for people living with HIV.

Healers are well positioned to address reported patient concerns, including: (1) keeping a patients HIV status a secret while providing support; (2) assisting with partner disclosure and initiating community/clinical systems of assistance if gender base violence is threatened/occurs; and (3) advocating for patients during clinical visits to ensure quality care is provided. Other programs in sub-Saharan Africa have shown that incorporating healers into an allopathic health system as adherence supporters for TB treatment is feasible, but healer use in HIV treatment is not well-documented. This novel intervention would provide patients newly initiated on ART a choice to nominate a specially trained healer as a treatment partner, and assess acceptability, feasibility, and patient outcomes using an interrupted time series quasi-experimental design. Community-based treatment partners can improve pharmacy adherence and loss to follow up , while decreasing stigma and isolation.

Engaging healers to conduct counseling sessions in a community setting to improve ART adherence necessitates technical clinical and psycho-social training. The ART Adherence Support Worker Training program will be adapted and used to train healers to be quality treatment partners and advocates. The training will ensure healers have the knowledge and skills to effectively: (1) Educate people living with HIV about treatment and HIV care; (2) Assess serious medication side effects or HIV co-infections; (3) Counsel patients about safer strategies for partner disclosure (with assistance if needed); (4) Accompany the patient for each clinical appointment; and (5) Advocate for quality health care delivery when assisting each patient. The training team will conduct training of the healers. All patients initiating treatment will be screened for interest in having a healer treatment partner. Control and intervention patients will be followed for one year, allowing the investigators to compare outcomes at 12-months to study the effectiveness of healers as adherence partners.

ELIGIBILITY:
Inclusion Criteria:

* Patients: Individuals 18 years of age or older, HIV-infected, and newly enrolled in ART and treatment services at Namacurra Sede.
* Traditional Healers: Healers will be eligible to participate if the healer lives within 10 km of the Namacurra Sede, received previous training from FGH, is 18 years of age or older, speak Portuguese, and see at least one patient per month

Exclusion Criteria:

* Patients: Individuals that are currently pregnant, HIV-uninfected, and/or not yet enrolled in HIV care. Individuals who cannot give consent due to mental limitations or intoxication.
* Traditional Healers: Healers who believe they can effectively treat or cure HIV or other associated conditions will be excluded from the project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Audet, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Namacurra Sede Health Facility, Namacurra, Zambezia Province, Mozambique

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Traditional Healer Support Program: This group will receive standard of care as described above plus support from a trained traditional healer.
  The intervention includes: (1) healer visits to the patient at home, healer support for couples counseling, healer provision of nutritional advice, and healer counsel about the importance of adherence. If anything is amiss, the healer will accompany the patient to the health facility for additional clinical services.
  Traditional Healer Support Program: Traditional Healers will provide the "traditional healer support program" assistance, as previously described, to all newly diagnosed patients.
  Standard of Care: First-line ART will consist of two nucleoside reverse-transcriptase inhibitors (NRTIs) plus a non-nucleoside reverse-transcriptase inhibitor (NNRTI)- TDF + 3TC (or FTC) + EFV as a fixed-dose combination to be taken twice a day for the rest of the patient's life), clinic-based counseling, and community searches if lost to follow up.
Period: Overall Study
Arm/Group | Standard of Care | Traditional Healer Support Program
Started | 170 | 150
Completed | 170 | 150
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Traditional Healer Support Program | Total
Number analyzed (Participants) | 170 | 150 | 320
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (11) | 33 (10) | 33 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 75 | 168
  Male | 77 | 75 | 152
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 170 | 150 | 320
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mozambique | 170 | 150 | 320
Employment [Count of Participants; unit: Participants] | 25 | 21 | 46

OUTCOME MEASURES:

1. Primary Outcome: Retention in Care
Description: We accessed the percentage of days where participants have medication. For example, if a participant picked up a 30 day supply of medication on August 1st but did not collect their next medication until October 1st, the patient would only be considered retained for 50% of the time.
Time Frame: Retention in care over 12 months
Population: Several patient ID numbers were not able to be matched to online database of patient records at this point give discrepancies in name or community. Given new paper records were introduced in 2019 we were not able to go back to the original records for cross-reference of medication pick-up.
Measure: Median (Inter-Quartile Range); unit: percentage of medication coverage
Groups:
- Standard of Care: This group will receive only standard of care HIV treatment, including ART medications (First-line ART will consist of two nucleoside reverse-transcriptase inhibitors (NRTIs) plus a non-nucleoside reverse-transcriptase inhibitor (NNRTI)- TDF + 3TC (or FTC) + EFV as a fixed-dose combination to be taken twice a day for the rest of the patient's life), clinic-based counseling, and community searches if lost to follow up.
  Standard of Care: First-line ART will consist of two nucleoside reverse-transcriptase inhibitors (NRTIs) plus a non-nucleoside reverse-transcriptase inhibitor (NNRTI)- TDF + 3TC (or FTC) + EFV as a fixed-dose combination to be taken twice a day for the rest of the patient's life), clinic-based counseling, and community searches if lost to follow up.
Arm/Group | Standard of Care | Traditional Healer Support Program
Number analyzed (Participants) | 163 | 113
percentage of medication coverage | 80 [48 to 92] | 79 [57 to 90]

2. Secondary Outcome: Viral Load
Description: Patient viral load at 12 months to assess the impact of the intervention on HIV viral suppression. HIV viral load tests are reported as the number of HIV copies in a milliliter (copies/mL) of blood using a reverse-transcriptase polymerase chain reaction (RT-PCR) test. If the viral load measurement is high, it generally indicates that HIV is present and replicating. Initial, untreated, and uncontrolled HIV viral loads can range as high as one million or more copies/mL. Viral loads that are consistently less than 200 copies/mL indicate that the virus is adequately suppressed and that the risk of disease progression is low. Viral load results below zero indicate that no virus was detected (this is how the outputs are recorded using the PRC test in the region. We did not assess change in values over time.
Time Frame: 12 months post-enrollment
Population: While this was one of our primary outcomes, less than 50% of our patients had a viral load within 2 months of the end of their first year in treatment. Laboratory capacity and transportation issues have been a problem in rural Mozambique for many years. While we were hoping this would be solved before the end of our study it was not.
Measure: Median (Inter-Quartile Range); unit: copies/mL
Groups:
- Traditional Healer Support Program: This group will receive standard of care as described above. In addition, the investigators will assess an intervention partnership with traditional healer including: community and clinic based support from a trained traditional healer.
  The intervention includes: (1) healer visits to the patient at home, healer support for couples counseling, healer provision of nutritional advice, and healer counsel about the importance of adherence. If anything is amiss, the healer will accompany the patient to the health facility for additional clinical services. In addition, the healer will accompany the patient on all regularly scheduled clinical visits.
  Traditional Healer Support Program: Traditional Healers will provide the "traditional healer support program" assistance, as previously described, to all newly diagnosed patients.
Arm/Group | Standard of Care | Traditional Healer Support Program
Number analyzed (Participants) | 75 | 37
copies/mL | -20 [-20 to 1326] | -20 [-20 to 1037]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Standard of Care | Traditional Healer Support Program
All-Cause Mortality (participants affected / at risk) | 14/170 | 15/150
Serious Adverse Events (participants affected / at risk) | 0/170 | 0/150
Other Adverse Events (participants affected / at risk) | 0/170 | 0/150

LIMITATIONS AND CAVEATS:
A pre-post intervention has inherent temporal biases. At the start of the intervention phase Mozambique shifted to a test-and-treat system; the patients in the post-intervention phase are likely substantively different from the pre-group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/59/NCT03076359/Prot_SAP_ICF_000.pdf